CLINICAL TRIAL: NCT03343197
Title: A Phase 1, Multicenter, Randomized, Controlled, Open-Label, Perioperative Study of AG-120 and AG-881 in Subjects With Recurrent, Non-Enhancing, IDH1 Mutant, Low Grade Glioma
Brief Title: Study of AG-120 and AG-881 in Subjects With Low Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG120-881-C-001
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Glioma
Keywords: Glioma; IDH1; AG-120; AG-881
MeSH Terms: conditions — Glioma | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- AG-120 (Experimental): AG-120 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle prior to surgery. Following surgery, subjects will have the option to receive treatment with AG-120 .
  Interventions: Drug: AG-120
- AG-881 (Experimental): AG-881 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle prior to surgery. Following surgery, subjects will have the option to receive treatment with AG-881.
  Interventions: Drug: AG881
- No Treatment Pre-Surgery (No Intervention): Subjects will not receive treatment prior to surgery. Following surgery, subjects will have the option to receive treatment with AG-120 or AG-881.

INTERVENTIONS:
Drug: AG-120 — Prior to surgery subjects will receive AG-120 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Subjects without residual disease following surgery will have the option to receive treatment for up to a year, until disease progression or unacceptable toxicity, whichever occurs first. Subjects with residual disease following surgery will have the option to receive treatment, until disease progression or unacceptable toxicity.
  Arms: AG-120
Drug: AG881 — Prior to surgery subjects will receive AG-881 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Subjects without residual disease following surgery will have the option to receive treatment for up to a year, until disease progression or unacceptable toxicity, whichever occurs first. Subjects with residual disease following surgery will have the option to receive treatment, until disease progression or unacceptable toxicity.
  Arms: AG-881

SUMMARY:
Study to evaluate the suppression of 2-HG (2-hydroxyglutarate) in IDH-1 mutant gliomas in resected tumor tissue following pre-surgical treatment with AG-120 or AG-881.

DETAILED DESCRIPTION:
A phase-1, multi-center study in recurrent non-enhancing gliomas with IDH1 R132H mutation for patients who require surgery. The purpose of this study is to evaluate the suppression of 2-HG by comparing the concentration of 2-HG in resected tumors from IDH1 mutant glioma subjects following AG-120 or AG-881 treatment with the 2-HG concentration in untreated, control tumors. The safety, tolerability, PK/PD, and anti tumor activity data from the study in subjects with recurrent non-enhancing Grade 2/3 LGG with an IDH1 R132H mutation for whom surgical resection is indicated will identify the recommended dose of AG-120 and AG-881 for future studies in glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age.
2. Have histologically or cytologically confirmed recurrent Grade 2 or 3 LGG (oligodendroglioma or astrocytoma according to World Health Organization 2016 classification).
3. Have documented IDH1 R132H gene mutation by local testing and known 1p19q or ATRX mutation status by local testing.
4. Have central confirmation of primarily non-enhancing disease by MRI with less than or equal to 5 mm slice thickness and up to 1 mm interslice gap on either 2D T2 weighted image, 3D T2 weighted image, or FLAIR, with at least 1 non-enhancing tumor measuring 1×1×1 cm.
5. Be candidates for clinical resection but for whom surgery is not urgently indicated (eg, for whom surgery within the next 2-4 months is appropriate).
6. Have KPS of ≥60%
7. Have expected survival of ≥12 months.

Exclusion Criteria:

1. Have received prior systemic anti-cancer therapy within 1 month of the first dose of AG-120 or AG-881 or have received an investigational agent <14 days prior to their first dose of AG-120 or AG-881. In addition, the first dose of AG-120 or AG-881 should not occur before a period of ≥5 half-lives of the investigational agent has elapsed.
2. Have had radiation within 6 months of the first dose of AG-120 or AG-881. (Note: Prior biopsy or surgery is allowed.)
3. Have received any prior treatment with an IDH inhibitor.
4. Have received any prior treatment with bevacizumab (Avastin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
2-HG concentration in surgically resected tumors | Up to 4 weeks, on average

SECONDARY OUTCOMES:
Safety and tolerability: incidence of adverse events and serious adverse events | Up to 48 weeks, on average
Pharmacodynamics of AG-120 or AG-881 measured by 2-HG concentration in plasma. | Up to 4 weeks, on average
Peak Plasma Concentration (Cmax) of AG-120 or AG-881 | Up to 4 weeks, on average
Time to maximum concentration (Tmax) of AG-120 or AG-881 | Up to 4 weeks, on average
Area Under the Curve (AUC) of AG-120 or AG-881 | Up to 4 weeks, on average
Elimination half-life of AG-120 or AG-881 | Up to 4 weeks, on average
Clinical activity associated with AG-120 or AG-881 according to modified RANO_LGG criteria. | Up to 48 weeks, on average

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - United States, California, Los Angeles, California
  - United States, California, San Francisco, California
  - United States, Massachusetts, Boston, Massachusetts
  - United States, New York, New York, New York
  - United States, North Carolina, Durham, North Carolina
  - United States, Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Mellinghoff IK, Lu M, Wen PY, Taylor JW, Maher EA, Arrillaga-Romany I, Peters KB, Ellingson BM, Rosenblum MK, Chun S, Le K, Tassinari A, Choe S, Toubouti Y, Schoenfeld S, Pandya SS, Hassan I, Steelman L, Clarke JL, Cloughesy TF. Vorasidenib and ivosidenib in IDH1-mutant low-grade glioma: a randomized, perioperative phase 1 trial. Nat Med. 2023 Mar;29(3):615-622. doi: 10.1038/s41591-022-02141-2. Epub 2023 Feb 23. PMID 36823302
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/